CLINICAL TRIAL: NCT03187977
Title: Cognitive Intervention at the End of Therapy for Survivors of Childhood ALL Treated on TOTXVI: A Pilot Study
Brief Title: Cognitive Intervention at the End of Therapy for Survivors of Childhood ALL Treated on TOTXVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ALLCOG; NCI-2017-01276 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Cognitive intervention; Survivors; Childhood ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the intervention group to receive cognitive training or to the standard of care group who will not receive cognitive training.
Who Masked: Outcomes Assessor
Masking Description: The study examiner (clinical research assistants or psychological examiners) will not know which group of participants is associated with each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training (Active Comparator): Participants will participate in computer-based cognitive training at the end of therapy.
  Interventions: Behavioral: Cognitive training
- Standard-of-Care (No Intervention): At the end of therapy, participants will participate in the current standard-of-care which does not include computer-based cognitive training.

INTERVENTIONS:
Behavioral: Cognitive training — Cogmed is a computer-based cognitive training program that consists of rotating exercises that train attention and working memory. The exercises are presented in a child-friendly, game-like format. The program is completed at home for 15-45 minutes each weekday for 5-9 weeks.
  Other Names: Cogmed
  Arms: Cognitive Training

SUMMARY:
Computer-based cognitive training has been found to be helpful for improving attention and working memory in pediatric and adult patients with existing cognitive difficulties. A previous study was conducted at St. Jude Children's Research Hospital with survivors of childhood cancer who were experiencing difficulties with attention and/or working memory. Findings from that study indicated that the use of Cogmed, computer-based cognitive training, is effective in improving attention and working memory in survivors.

Researchers want to learn whether Cogmed intervention completed at the end of therapy for acute lymphoblastic leukemia will be effective for all survivors (i.e., regardless of whether they have existing difficulties).

PRIMARY OBJECTIVES:

* To evaluate the overall participation rate in a randomized, standard-of-care controlled trial of computerized cognitive intervention administered at the end of TOTXVI therapy.
* To estimate the study completion rate in a randomized, standard-of-care controlled trial of computerized cognitive intervention administered at the end of TOTXVI therapy.
* To estimate the compliance rate for participants randomized to the intervention arm of a computerized cognitive intervention administered at the end of TOTXVI therapy.
* To estimate the standard deviation for the overall cohort on a measure of working memory.
* To use neuroimaging data collected in the context of the Total Therapy XVI trial to explore candidate biomarkers predictive of response to the computerized cognitive intervention.

DETAILED DESCRIPTION:
Participants enrolled on the TOTXVI protocol at SJCRH will be randomized to either complete the Cogmed intervention at the end of their therapy, or to a standard-of-care condition.

Cogmed is a computer-based cognitive training program that consists of rotating exercises that train attention and working memory. The exercises are presented in a child-friendly, game-like format. Training is completed at home in 25 sessions for 15-45 minutes each weekday for 5-9 weeks. A research team member serves as a coach who monitors progress and provides support through weekly phone calls with study participants and their parents/guardians. Information regarding compliance and performance is tracked over the internet and used to tailor feedback during weekly telephone coaching.

Neurocognitive assessments will be conducted at baseline, immediate-post (3-4 months after baseline), and 8 month follow-up (12 months after baseline).

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled and receiving treatment for acute lymphoblastic leukemia (ALL) on the TOTXVI therapy protocol at St. Jude Children's Research Hospital
* At least 4 years of age at the time of randomization
* Primary language is English
* Parent/legal guardian/caregiver that speaks English available to assist in participant's training

Exclusion Criteria:

* Significant cognitive impairment as determined by either an IQ of ≤ 70 or by clinician judgment
* Major sensory or motor impairment that would preclude valid cognitive testing
* Major psychological condition that would preclude completion of the intervention
* History of significant CNS injury or disease predating or unrelated to cancer diagnosis
* Documented ADHD predating cancer diagnosis

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Change in working memory | Prior to intervention (baseline) and post intervention (up to one year later)
  The magnitude and standard deviation of pre- to post-change in Spatial Span Backward will be estimated for each group and for the overall group.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M. Jacola, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://stjude.org
- See also: Clinical Trials Open at St. Jude — http://stjude.org/protocols